CLINICAL TRIAL: NCT07249437
Title: Non-invasive Methods for Oral Cancer Screening
Acronym: HRME
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 202503081RINA
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Oral Cancer Screening
Keywords: oral cancer; high-resolution microendoscopy (HRME)
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — plasma serum buffy-coat+RBC Liquid-Based Cytology，LBC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oral cancer is a common cancer worldwide, with approximately 250,000 new cases annually and a high mortality rate. Its major risk factors include smoking, alcohol consumption, and betel nut chewing. Current screening methods rely heavily on visual inspection by specialist physicians and invasive biopsy of lesions, but they suffer from limitations such as insufficient sensitivity, sampling errors in biopsies, and low patient compliance.

This study proposes an innovative cross-sectional randomized trial aimed at evaluating two non-invasive techniques-oral digital imaging photography (high-resolution microendoscopy, HRME) and liquid-based cytology (LBC) of the oral mucosa-in order to optimize the screening of oral precancerous lesions.

DETAILED DESCRIPTION:
Oral cancer is a common malignancy worldwide, with approximately 250,000 new cases diagnosed annually and a high mortality rate. Its primary risk factors are smoking, alcohol consumption, and betel nut chewing. Current screening methods heavily rely on visual inspection by specialist physicians and invasive biopsy of lesions, but they are limited by insufficient sensitivity, biopsy sampling errors, and low patient compliance.

To address these issues, this study proposes an innovative cross-sectional randomized trial to evaluate two non-invasive techniques-high-resolution microendoscopy (HRME) and liquid-based cytology (LBC) of the oral mucosa-with the aim of optimizing screening for oral precancerous lesions.

The study will recruit 400 participants with visually identified oral potentially malignant disorders (e.g., leukoplakia or erythroplakia) and randomly assign them to two groups:

a clinical biopsy group (biopsy site selected based on conventional visual inspection), and an HRME-guided biopsy group (biopsy site directed by high-resolution microendoscopy).

Both groups will also undergo liquid-based cytology (LBC) through collection and analysis of oral mucosal cells.

The study objectives include:

Comparing the detection rates of precancerous lesions (mild, moderate, severe dysplasia, or carcinoma in situ, or invasive cancer) between the two groups; Analyzing the intra-lesional consistency of biopsy sites in both groups; Validating the diagnostic performance of LBC alone or in combination with HRME.

ELIGIBILITY:
Inclusion Criteria:We proposed to include individuals aged 30-80 years with prevalent oral precancer with or without a prior history of head and neck cancer (oral cavity, oropharynx, hypopharynx, larynx). The rationale for including those with history of cancer is that they are still at risk of developing oral cavity cancer and therefore will benefit from a better screening algorithm. Also, in our experience lesions in cancer survivors are phenotypically similar to those without a prior history of head and neck cancer. Only lesions with at least 1 cm in greatest diameter will be considered eligible. Additionally, because there could be issues in HRME imaging due to keratinization at some anatomic sites, we will divide lesions into approximate quadrants and exclude any lesions that do not have good nuclear resolution on at least one representative image per quadrant.

-

Exclusion Criteria:We exclude those who: 1) are undergoing current cancer treatment or had a cancer within the last two years to avoid any effects of the cancer treatments; 2) are unwilling or unable to provide informed consent to participate; and/or 3) based on clinical judgement, should not be included in the study e.g., has other medical conditions that would preclude them from participating.

-

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We proposed to include individuals aged 30-80 years with prevalent oral precancer with or without a prior history of head and neck cancer (oral cavity, oropharynx, hypopharynx, larynx).
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Whether the biopsy sites are consistent | one month
  Whether the biopsy site selected based on conventional physician visual inspection is the same area as the biopsy site selected with the assistance of oral digital imaging (high-resolution microendoscopy, HRME) each time.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Ping Wang, Doctor, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
For the needs of this research, the specimens we collect from you will be used in accordance with this research protocol. The specimens will be stored either in the laboratory of Dr. Cheng-Ping Wang at National Taiwan University Hospital or at the U.S. National Institutes of Health (NIH) and will be retained for a maximum of 30 years. Upon expiration of the 30-year storage period, the specimens will be destroyed in accordance with the law.
  To protect your personal privacy, your name and other personally identifiable information will be replaced with a unique study/research ID number, ensuring that your specimens and related data remain completely confidential.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2027/4/30~2057/4/30
Access Criteria: DCEG, NCI Investigator(s): Anil K. Chaturvedi and Philip E. Castle U.S. Co-Investigator(s): Kelly J. Yu (IIB), Hormuzd A. Katki (BB), Li C. Cheung (BB), Maria Demarco (CGB), Mark W. Lingen (University of Chicago), Abberly Lott-Limbach (Ohio State University), Ann Gillenwater (MD Anderson), Rebecca Richards-Kortum (Rice University), Richard Schwarz (Rice University), Nadarajah Vigneswaran (UTHealth School of Dentistry at Houston), and Jennifer Carns Plante (Rice University).
  Taiwan Co-Investigator(s): Tseng-Cheng Chen (National Taiwan University Hospital), Pei-Jen Lou (National Taiwan University Hospital), Yu-Fong Chang (National Taiwan University Hospital),Min-Shu Hsieh (National Taiwan University Hospital), Chun-Yang Hung(National Taiwan University Hospital) ,and Cheng-Ping Wang (National Taiwan University Hospital)